CLINICAL TRIAL: NCT02729688
Title: Effectiveness of a Pressure Indicator Guided and a Conventional Bandaging in Treatment of Venous Leg Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRIRAJ016/2559
Record Dates: First submitted 2016-03-25; First posted 2016-04-06 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Venous Insufficiency
Keywords: Venous insufficiency; Compression; Bandaging
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ordinary elastic bandage (Active Comparator): Bandaging was applied by spiral methods. Three ordinary elastic bandages were applied with 50 % stretching and 50% overlapping from foot to just below knee level.
  Interventions: Device: Ordinary elastic bandage
- customized pressure guide bandage (Active Comparator): Bandaging was applied by spiral methods. Three customized pressure guide elastic bandage were applied by stretching until the elliptical shape marker in the bandage turned into circular shape with 50% overlapping from foot to just below knee level.
  Interventions: Device: customized pressure guide bandage

INTERVENTIONS:
Device: customized pressure guide bandage — Investigators developed the customized pressure guide elastic bandage (CPG-EB). The experienced nurse applied the elastic bandages to each patient with sub bandage pressure monitoring. The target pressure was 35-45 mmHg. Measurements of the pressure applied by bandages was performed at point B1 corresponding to the height where the Achilles' tendon turns into the gastrocnemius muscle with Picopress (MicroLAB Elettronica, Ponte S. Nicolo, Italy). If the target pressure 35-45 mmHg was achieved, the circular ink stamp was applied into the entire bandages. The markers in CPG-EB had elliptical shape when they were not stretched. They turned into circular shape when they were stretched.
  For the OEB, Bandaging was applied by spiral methods. Three EB were applied with 50 % stretching and 50% overlapping from foot to just below knee level.
  Arms: customized pressure guide bandage
Device: Ordinary elastic bandage — Bandaging was applied by spiral methods. Three ordinary elastic bandages were applied with 50 % stretching and 50% overlapping from foot to just below knee level.
  Arms: ordinary elastic bandage

SUMMARY:
Objective of this study are to compare the interface pressure by applying ordinary elastic bandage (OEB) and CPG-EB. In addition, investigators compared the percentage of patients who could apply the optimal pressure with OEB and CPG-EB.

DETAILED DESCRIPTION:
For treatment of venous ulcer, it was shown that compression bandaging of 35-45 mmHg sub-bandage pressure at the ankle was shown in several studies to be safe and effective.The efficacy of compression bandage considerably depends on the applied pressure and it is therefore largely dependent on the individual applying bandages. The lower pressure leads to treatment failure while the higher pressure leads to skin complication.

The use of objective devices to proof that the bandage is sufficiently applied is not available for every patients. To help the patients to apply the bandage with optimal pressure, investigators developed the customized pressure guide elastic bandage (CPG-EB) by using sub-bandage pressure guidance.

Objective of this study are to compare the interface pressure by applying ordinary elastic bandage (OEB) and CPG-EB. In addition,investigators compared the percentage of inexperienced staffs who could apply the optimal pressure with OEB and CPG-EB.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic venous insufficiency CEAP (clinical, etiologic, anatomic, and pathophysiologic) C4,C5 and C6

Exclusion Criteria:

* Patients who can not perform bandaging by themselves

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Sub-bandage pressure | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Nuttawut Sermsathanasawadi, MD, Principal Investigator — Mahidol University
Locations (1):
- Vascular Surgery, Siriraj Hospital, Mahidol University, Bangkoknoi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sermsathanasawadi N, Tarapongpun T, Pianchareonsin R, Puangpunngam N, Wongwanit C, Chinsakchai K, Mutirangura P, Ruangsetakit C. Customizing elastic pressure bandages for reuse to a predetermined, sub-bandage pressure: A randomized controlled trial. Phlebology. 2018 Oct;33(9):627-635. doi: 10.1177/0268355517746434. Epub 2017 Dec 25. PMID 29277134